CLINICAL TRIAL: NCT05296798
Title: A Phase III, Randomized, Open-Label Study Evaluating the Efficacy and Safety of Giredestrant in Combination With Phesgo Versus Phesgo After Induction Therapy With Phesgo + Taxane in Patients With Previously Untreated HER2-Positive, Estrogen Receptor-Positive Locally-Advanced or Metastatic Breast Cancer
Brief Title: A Study to Evaluate the Efficacy and Safety of Giredestrant in Combination With Phesgo (Pertuzumab, Trastuzumab, and Hyaluronidase-zzxf) Versus Phesgo in Participants With Locally Advanced or Metastatic Breast Cancer (heredERA Breast Cancer)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WO43571; 2022-500014-26-00 (Registry Identifier: EU Clinical Trials)
Record Dates: First submitted 2022-03-23; First posted 2022-03-25 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced or Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab; Trastuzumab; Injections, Subcutaneous; giredestrant; Docetaxel; Paclitaxel; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Induction Therapy: Phesgo plus Taxane-Based Chemotherapy (Other)
  Interventions: Drug: Phesgo; Drug: Docetaxel; Drug: Paclitaxel
- Arm A, Maintenance Therapy: Phesgo (Active Comparator)
  Interventions: Drug: Phesgo; Drug: LHRH Agonist; Drug: Optional Endocrine Therapy of Investigator's Choice
- Arm B, Maintenance Therapy: Giredestrant plus Phesgo (Experimental)
  Interventions: Drug: Phesgo; Drug: Giredestrant; Drug: LHRH Agonist

INTERVENTIONS:
Drug: Phesgo — Phesgo will be administered subcutaneously (SC) at a fixed non-weight-based dose. In the induction therapy phase, a loading dose (1200 milligram (mg) pertuzumab, 600 mg trastuzumab, and 30,000 units of recombinant human PH20 hyaluronidase [rHuPH20]) will be administered in the first cycle (1 cycle is 21 days). In subsequent cycles, maintenance doses (600 mg pertuzumab, 600 mg trastuzumab, and 20,000 units rHuPH20) will be administered once every 3 weeks (Q3W).
  Other Names: Pertuzumab, Trastuzumab, and Hyaluronidase-zzxf; Pertuzumab, Trastuzumab, and rHuPH20; Fixed-Dose Combination of Pertuzumab and Trastuzumab for Subcutaneous Use (PH FDC SC); RO7198574; RG6264
Drug: Giredestrant — A 30 milligram (mg) capsule of giredestrant will be taken orally once a day on Days 1 to 21 of each 21-day cycle.
  Other Names: GDC-9545; RO7197597; RG6171
  Arms: Arm B, Maintenance Therapy: Giredestrant plus Phesgo
Drug: Docetaxel — During the induction therapy phase, the investigator's choice of taxane-based chemotherapy (i.e., docetaxel or paclitaxel) will be administered after Phesgo. Docetaxel will be administered at 75 milligrams per metre squared of body surface area (mg/m2) intravenously over 60 (±10) minutes on Day 1 of each cycle for 4 to 8 cycles (a cycle is 21 days); this dose may be escalated to 100 mg/m2 if the initial dose was well tolerated.
  Arms: Induction Therapy: Phesgo plus Taxane-Based Chemotherapy
Drug: Paclitaxel — During the induction therapy phase, the investigator's choice of taxane-based chemotherapy (i.e., docetaxel or paclitaxel) will be administered after Phesgo. Paclitaxel will be administered at 80 milligrams per metre squared of body surface area (mg/m2) intravenously over a minimum of 1 hour on Days 1, 8, and 15 of each cycle for 4 to 8 cycles (a cycle is 21 days); this weekly regimen is considered as one complete cycle whenever 3 weekly doses are given.
  Arms: Induction Therapy: Phesgo plus Taxane-Based Chemotherapy
Drug: LHRH Agonist — A luteinizing hormone-releasing hormone (LHRH) agonist will be administered every 28 days to pre- and peri-menopausal women and all male participants while receiving giredestrant in Arm B. An LHRH agonist may be administered to male participants and pre- and peri-menopausal female participants receiving tamoxifen in Arm A, and should be administered to those receiving an aromatase inhibitor in Arm A. The investigator will determine and supply the appropriate LHRH agonist locally approved for use in breast cancer. The LHRH agonist will be administered according to local prescribing information.
  Arms: Arm A, Maintenance Therapy: Phesgo; Arm B, Maintenance Therapy: Giredestrant plus Phesgo
Drug: Optional Endocrine Therapy of Investigator's Choice — For participants in Arm A, optional endocrine therapy of investigator's choice is allowed based on the standard of care, and it can include an aromatase inhibitor or tamoxifen with or without an LHRH agonist, or gonadal ablation. The decision to include or exclude this option must be made prior to randomization.
  Arms: Arm A, Maintenance Therapy: Phesgo

SUMMARY:
This Phase III, randomized, two-arm, open-label, multicenter study will evaluate the efficacy and safety of giredestrant plus Phesgo compared with Phesgo after induction therapy with Phesgo plus taxane in participants with human epidermal growth factor receptor 2 (HER2)-positive, estrogen receptor (ER)-positive advanced breast cancer (metastatic or locally advanced disease not amenable to curative treatment) who have not previously received a systemic non-hormonal anti-cancer therapy in the advanced setting.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed and documented human epidermal growth factor receptor 2 (HER2)-positive/estrogen receptor (ER)-positive adenocarcinoma of the breast with metastatic or locally-advanced disease not amenable to curative resection
* At least one measurable lesion and/or non-measurable disease evaluable according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Disease-free interval from completion of adjuvant or neoadjuvant systemic non-hormonal treatment to recurrence of ≥6 months
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
* Left ventricular ejection fraction (LVEF) of at least (≥)50% measured by echocardiogram (ECHO) or multiple-gated acquisition scan (MUGA)
* Adequate hematologic and end-organ function
* For women of childbearing potential: Participants who agree to remain abstinent (refrain from heterosexual intercourse) or use contraception, and agree to refrain from donating eggs, during the treatment period and for 7 months after the final dose of Phesgo
* For men: participants who agree to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agree to refrain from donating sperm, during the treatment period and for 7 months after the final dose of Phesgo to avoid exposing the embryo

Maintenance Phase Inclusion Criteria

* Complete a minimum of four cycles to a maximum of eight cycles of induction therapy; the minimum cycles are defined as either: Phesgo injections + 4 docetaxel infusions, or Phesgo injections + 12 paclitaxel infusions
* Achieve a minimum of stable disease (SD) (or Non-complete response [CR]/Non-progressive disease [PD] for participants with non-measurable disease) (i.e., did not experience PD) according to RECIST v1.1 at the last tumor assessment during the induction therapy phase
* LVEF of ≥50% at the last assessment during the induction therapy phase

Exclusion Criteria:

* Previous systemic non-hormonal anti-cancer therapy in the metastatic breast cancer (MBC) or advanced breast cancer (ABC) setting. Note: Up to one line of single-agent endocrine therapy given in the metastatic or locally advanced setting will be allowed.
* Prior treatment with a selective estrogen receptor degrader (SERD)
* Previous treatment with approved or investigative anti-HER2 agents in any breast cancer treatment setting, except Phesgo (or trastuzumab SC with pertuzumab IV, or pertuzumab and trastuzumab IV), single-agent trastuzumab IV or SC, ado-trastuzumab emtansine, lapatinib, and neratinib in the neoadjuvant or adjuvant setting
* Disease progression within 6 months of receiving adjuvant anti-HER2 therapy (such as trastuzumab, with or without pertuzumab [IV, SC, or fixed-dose combination], or ado-trastuzumab emtansine, or neratinib)
* Non-resolution of all acute toxic effects of prior anti-cancer therapy or surgical procedures to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE v5.0) Grade 1 or better
* History of persistent Grade ≥2 (NCI-CTC, Version 5.0) hematological toxicity resulting from previous adjuvant or neo-adjuvant therapy
* History of exposure to the following cumulative doses of anthracyclines; Doxorubicin >360 mg/m2; Liposomal doxorubicin >500 mg/m2; Epirubucin >720 mg/m2; Mitoxantrone >120 mg/m2; Idarubicin >90 mg/m2.
* Known active uncontrolled or symptomatic central nervous system (CNS) metastases, carcinomatous meningitis, or leptomeningeal disease
* Dyspnea at rest due to complications of advanced malignancy, or other disease requiring continuous oxygen therapy
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 7 months after the final dose of Phesgo (Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of induction therapy).
* Treated with investigational therapy within 28 days prior to initiation of induction therapy
* Treated with localized palliative radiotherapy within 14 days prior to initiation of induction therapy
* Concurrent participation in any other therapeutic clinical trial
* Known hypersensitivity to any of the study medications or to excipients of recombinant human or humanized antibodies
* Current chronic daily treatment (continuous for >3 months) with corticosteroids (dose of 10 mg/day methylprednisolone or equivalent)
* Poorly controlled hypertension
* Known clinically significant history of liver disease consistent with Child-Pugh Class B or C, active liver disease including active viral or other hepatitis virus, autoimmune hepatic disorders, or sclerosing cholangitis, current alcohol abuse, or cirrhosis
* Active cardiac disease or history of cardiac dysfunction
* Major surgical procedure or significant traumatic injury within 14 days prior to enrollment or anticipation of need for major surgery during induction therapy
* Active inflammatory bowel disease, chronic diarrhea, short bowel syndrome, or major upper gastrointestinal surgery
* Concurrent, serious, uncontrolled infections, or known infection with HIV with the following exception: Individuals who are HIV positive are eligible provided they are stable on anti-retroviral therapy for ≥4 weeks, have a CD4 count ≥350 cells/uL, and have an undetectable viral load and no history of AIDS-defining opportunistic infections within 12 months prior to enrollment.
* Serious COVID-19 infection within 14 days prior to enrollment; however, no screening testing for SARS-CoV-2 is required
* Serious infection requiring oral or IV antibiotics within 7 days prior to screening
* Any serious medical condition or abnormality in clinical laboratory tests that precludes an individual's safe participation in the study
* History of malignancy within 5 years prior to screening with the exception of the cancer under investigation in this study and malignancies with a negligible risk of metastasis or death
* For pre- and perimenopausal women, and men: Known hypersensitivity to luteinizing hormone-releasing hormone agonist (LHRHa); Not willing to undergo and maintain treatment with approved LHRHa therapy for the duration of endocrine therapy that requires gonadal function suppression
* Treatment with strong CYP3A4 inhibitors or inducers within 14 days or 5 drug-elimination half-lives, whichever is longer, prior to initiation of giredestrant treatment in Arm B
* A documented history of hemorrhagic diathesis, coagulopathy, or thromboembolism, including deep vein thrombosis, unless the condition is adequately treated and under control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 922 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival, as Determined by the Investigator According to RECIST v1.1 | From randomization for maintenance therapy to the first occurrence of disease progression or death from any cause, whichever occurs first (up to 53 months)

SECONDARY OUTCOMES:
Overall Survival | From randomization for maintenance therapy to death from any cause (up to 98 months)
Objective Response Rate, as Determined by the Investigator According to RECIST v1.1 | From randomization for maintenance therapy to disease progression or death (up to 53 months)
  The objective response rate is defined as the percentage of participants with a complete response (CR) or partial response (PR) on two consecutive occasions at least 4 weeks apart.
Duration of Response, as Determined by the Investigator According to RECIST v1.1 | From first occurrence of documented objective response after randomization for maintenance therapy to disease progression or death from any cause, whichever occurs first (up to 53 months)
Clinical Benefit Rate, as Determined by the Investigator According to RECIST v1.1 | From randomization for maintenance therapy to disease progression or death (up to 53 months)
  The clinical benefit rate is defined as the percentage of participants with stable disease for ≥24 weeks or a complete response (CR) or partial response (PR).
Mean Role Functioning Score Over Time, as Assessed Using the European Organisation for Research and Treatment of Cancer Quality of Life-Core 30 (EORTC QLQ-C30) Questionnaire | Maintenance Cycles 1 (Baseline), 3, 6, 9, 12, 15, 18, once every 6 cycles from Cycles 24 to 90 (1 cycle is 21 days), treatment discontinuation, every 6 months and every year for Follow-up Years 1-2 and 3-5, respectively (up to 8 years)
Mean Change from Baseline in the Role Functioning Score Over Time, as Assessed Using the European Organisation for Research and Treatment of Cancer Quality of Life-Core 30 (EORTC QLQ-C30) Questionnaire | Maintenance Cycles 1 (Baseline), 3, 6, 9, 12, 15, 18, once every 6 cycles from Cycles 24 to 90 (1 cycle is 21 days), treatment discontinuation, every 6 months and every year for Follow-up Years 1-2 and 3-5, respectively (up to 8 years)
Mean Physical Functioning Score Over Time, as Assessed Using the European Organisation for Research and Treatment of Cancer Quality of Life-Core 30 (EORTC QLQ-C30) Questionnaire | Maintenance Cycles 1 (Baseline), 3, 6, 9, 12, 15, 18, once every 6 cycles from Cycles 24 to 90 (1 cycle is 21 days), treatment discontinuation, every 6 months and every year for Follow-up Years 1-2 and 3-5, respectively (up to 8 years)
Mean Change from Baseline in the Physical Functioning Score Over Time, as Assessed Using the European Organisation for Research and Treatment of Cancer Quality of Life-Core 30 (EORTC QLQ-C30) Questionnaire | Maintenance Cycles 1 (Baseline), 3, 6, 9, 12, 15, 18, once every 6 cycles from Cycles 24 to 90 (1 cycle is 21 days), treatment discontinuation, every 6 months and every year for Follow-up Years 1-2 and 3-5, respectively (up to 8 years)
Mean Global Health Status/Quality of Life Score Over Time, as Assessed Using the European Organisation for Research and Treatment of Cancer Quality of Life-Core 30 (EORTC QLQ-C30) Questionnaire | Maintenance Cycles 1 (Baseline), 3, 6, 9, 12, 15, 18, once every 6 cycles from Cycles 24 to 90 (1 cycle is 21 days), treatment discontinuation, every 6 months and every year for Follow-up Years 1-2 and 3-5, respectively (up to 8 years)
Mean Change from Baseline in the Global Health Status/Quality of Life Score Over Time, as Assessed Using the European Organisation for Research and Treatment of Cancer Quality of Life-Core 30 (EORTC QLQ-C30) Questionnaire | Maintenance Cycles 1 (Baseline), 3, 6, 9, 12, 15, 18, once every 6 cycles from Cycles 24 to 90 (1 cycle is 21 days), treatment discontinuation, every 6 months and every year for Follow-up Years 1-2 and 3-5, respectively (up to 8 years)
Number of Participants with at Least One Adverse Event, with Severity Determined According to National Cancer Institute Common Terminology Criteria for Adverse Events, version 5 (NCI CTCAE v5.0) | From Baseline until 28 days after the final dose of study treatment (up to 8 years, 5 months)
Number of Participants with Abnormalities in Clinical Laboratory Test Results | From Baseline until 28 days after the final dose of study treatment (up to 8 years, 5 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (208):
- United States (18):
  - Arizona Clinical Research Center, Inc, Tucson, Arizona
  - Los Angeles Hematology Oncology Medical Group, Los Angeles, California
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Carle Cancer Center, Urbana, Illinois
  - Maryland Oncology Hematology - Annapolis, Annapolis, Maryland
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Queens Hospital Cancer Center, Jamaica, New York
  - Clinical Research Alliance, Westbury, New York
  - West Cancer Center, Germantown, Tennessee
  - CHRISTUS Spohn Cancer Center - Shoreline, Corpus Christi, Texas
  - Texas Oncology - DFW, Dallas, Texas
  - Texas Oncology - El Paso, El Paso, Texas
  - CHRISTUS St. Michael Health System, Texarkana, Texas
  - Swedish Cancer Institute - Edmonds Campus, Edmonds, Washington
  - Swedish Cancer Institute - Issaquah, Issaquah, Washington
  - Swedish Cancer Institute, Seattle, Washington
- Argentina (7):
  - Centro de Investigaciones Médicas y Desarrollo LC S.R.L, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Centro Oncologico Korben, Ciudad Autonoma Buenos Aires
  - Centro Oncologico Riojano Integral (CORI), La Rioja
  - Fundacion Centro Oncologico de Integracion Regional (COIR), Mendoza
  - Instituto de Oncología de Rosario, Rosario
  - Hospital Provincial del Centenario, Rosario
  - CER San Juan Centro Polivalente de Asistencia e Investigacion Clinica, San Juan
- Belgium (5):
  - GHdC Site Les Viviers, Charleroi
  - UZ Gent, Ghent
  - Jessa Zkh (Campus Virga Jesse), Hasselt
  - UZ Leuven Gasthuisberg, Leuven
  - Clinique Ste-Elisabeth, Namur
- Brazil (10):
  - Pronutrir - suporte nutricional e quimioterapia ltda., Fortaleza, Ceará
  - Hospital Sao Rafael - HSR, Salvador, Estado de Bahia
  - Hospital Araujo Jorge, Goiânia, Goiás
  - Hospital do Câncer de Londrina, Londrina, Paraná
  - Hospital do Cancer de Pernambuco - HCP, Recife, Pernambuco
  - Oncosite - Centro de Pesquisa Clinica Em Oncologia Ltda, Ijuí, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Hospital de Amor Amazônia, Porto Velho, Rondônia
  - Fundação Pio XII Hospital de Câncer de Barretos, Barretos, São Paulo
  - Clinica de Pesquisa e Centro de Estudos em Oncologia Ginecologica e Mamaria Ltda, São Paulo, São Paulo
- China (23):
  - Affiliated Hospital of Hebei University, Baoding
  - Peking University People's Hospital, Beijing
  - the First Affiliated Hospital of Bengbu Medical College, Bengbu
  - The First Hospital of Jilin University, Changchun
  - Hunan Cancer Hospital, Changsha
  - Sichuan Cancer Hospital, Chengdu
  - West China Hospital - Sichuan University, Chengdu
  - No. 900 Hospital (Fuzhou General Hospital), Fuzhou
  - Fujian Cancer Hospital, Fuzhou
  - Zhejiang Provincial People?s Hospital, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Shandong Cancer Hospital, Jinan
  - The First Affiliated Hospital Of Jinzhou Medical University, Jinzhou
  - Yunnan Cancer Hospital, Kunming
  - Jiangxi Cancer Hospital, Nanchang
  - Jiangsu Cancer Hospital, Nanjing
  - Jiangsu Province Hospital (the First Affiliated Hospital With Nanjing Medical University), Nanjing
  - Guangxi Cancer Hospital of Guangxi Medical University, Nanning
  - The First Affiliated Hospital of China Medical University, Shenyang
  - Tianjin Cancer Hospital, Tianjin
  - The Tumor Hospital of Xinjiang Medical University, Ürümqi
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xian Jiao Tong University, Xi'an
- Colombia (4):
  - Fundación CTIC - Centro de Tratamiento e Investigación sobre Cáncer Luis Carlos Sarmiento Angulo, Bogota, D.C.
  - Clinica Colsanitas S.A. sede Clinica Universitaria Colombia, Bogotá
  - Oncomedica S.A., Montería
  - Oncólogos de Occidente, Pereira
- Egypt (3):
  - Dar El salam Cancer Centre, Cairo
  - National Cancer Institute- Breast Cancer Treatment & Research Hospital - 5th settlement, Cairo
  - Sohag Oncology Center, Cairo
- France (9):
  - Institut Sainte Catherine, Avignon
  - CH de la Côte Basque - Hôpital de Bayonne, Bayonne
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - CHU de GRENOBLE, Grenoble
  - CHD Vendée, La Roche-sur-Yon
  - Hopital Prive Jean Mermoz, Lyon
  - INSTITUT CURIE_Site Paris, Paris
  - Centre Catalan D' Oncologie, Perpignan
- Germany (14):
  - Gesundheitszentrum Wetterau, Hochwaldkrankenhaus Bad Nauheim, Bad Nauheim
  - Sozialstiftung Bamberg, Klinikum am Bruderwald, Gynäkologie, Bamberg
  - Gynäkologisches Zentrum Bonn, Bonn
  - Onkozentrum Dres. Göhler, Dresden
  - Kliniken Essen-Mitte, Essen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Nationales Centrum für Tumorerkrankungen (NCT), Heidelberg
  - Ärztehaus am Bahnhofsplatz, Hildesheim
  - Universitätsklinikum des Saarlandes, Homburg/Saar
  - Dres. Andreas Köhler und Roswitha Fuchs, Langen
  - MVZ für Hämatologie und Onkologie Ravensburg GmBH, Ravensburg
  - Caritas-Krankenhaus St. Josef, Regensburg
  - Klinikum Mutterhaus der Borromaeerinnen gGmbH, Trier
  - Universitätsklinik Tübingen, Tübingen
- Hungary (6):
  - Budapesti Szent Margit Korhaz, Budapest
  - Semmelweis Egyetem;Onkológiai Profil (Belgyógyászati és Onkológiai Klinika), Budapest
  - Bekes Varmegyei Központi Korhaz, Pandy Kalman Tagkorhaz, Gyula
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz-Rendelointezet, Szolnok
  - Komarom-Eszergom Varmegyei Szent Borbala Korhaz, Tatabánya
- India (7):
  - Manipal Hospital, Bangalore, Karnataka
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - Sahyadri Super Specialty Hospital Hadapsar, Pune, Maharashtra
  - Rajiv Gandhi Cancer Inst.&Research Center, New Delhi, National Capital Territory of Delhi
  - Fortis Hospital, New Delhi, National Capital Territory of Delhi
  - Netaji Subhas Chandra Bose Cancer Hospital, Kolkata, West Bengal
  - TATA Medical Centre, Kolkata, West Bengal
- Italy (11):
  - Azienda Ospedaliera Universitaria Federico II, Napoli, Campania
  - Istituto Nazionale Tumori Irccs Fondazione g. PASCALE, Napoli, Campania
  - Azienda Unità Sanitaria Locale di Reggio Emilia/IRCCS, Reggio Emilia, Emilia-Romagna
  - Ospedale Infermi AUSL della Romagna, Rimini, Emilia-Romagna
  - Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - Asst Degli Spedali Civili Di Brescia, Brescia, Lombardy
  - Istituto Europeo Di Oncologia, Milan, Lombardy
  - Istituto Clinico Humanitas, Rozzano, Lombardy
  - Humanitas Centro Catanese Di Oncologia, Misterbianco (CT), Sicily
  - Ospedale Civile, Livorno, Tuscany
  - IOV - Istituto Oncologico Veneto - IRCCS, Padua, Veneto
- King Hussein Cancer Center, Amman, Jordan
- Kenya (2):
  - International Cancer Institute (ICI), Eldoret
  - The Aga Khan University-Kenya., Nairobi
- Lebanon (2):
  - Rizk Hospital, Beirut
  - American University of Beirut - Medical Center, Beirut
- Mexico (10):
  - Investigacion Oncofarmaceutica, La Paz, Baja California Sur
  - Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco
  - Iem-Fucam, D.F., Mexico CITY (federal District)
  - Health Pharma Professional Research, Mexico City, Mexico CITY (federal District)
  - Filios Alta Medicina, Monterrey, Nuevo León
  - Hospital Universitario, Monterrey, Nuevo León
  - Hospital Zambrano Hellion TecSalud, Monterrey, Nuevo León
  - Cuidados oncologicos, Querétaro City, Querétaro
  - Oncologico Potosino, San Luis Potosí City, San Luis Potosí
  - Centro Estatal de Cancerologia de Chihuahua, Chihuahua City
- Sultan Qaboos Comprehensive Cancer Care & Research Center, Muscat, Oman
- Poland (8):
  - Uniwersyteckie Centrum Kliniczne, Klinika Onkologii i Radioterapii, Gdansk
  - Przychodnia Lekarska KOMED, Roman Karaszewski, Konin
  - Szpital Wojewódzki im. Miko?aja Kopernika, Koszalin
  - Opolskie Centrum Onkologii, Opole
  - Ars Medical Sp. z o. o., Pi?a
  - Szpital Kliniczny im. H.Swiecickiego UM w Poznaniu, Późna
  - MRUKMED Lekarz Beata Madej-Mruk i Partner Spolka Partnerska Oddzial nr 1 w Rzeszowie, Rzeszów
  - Centrum Onkologii ? Instytut im. Marii Sk?odowskiej-Curie Klinika Nowotworów Piersi i Chirurgii, Warsaw
- Portugal (4):
  - IPO de Coimbra, Coimbra
  - Hospital de S. Francisco Xavier, Lisbon
  - Hospital Beatriz Angelo, Loures
  - IPO do Porto, Porto
- Saudi Arabia (3):
  - King Faisal Specialist Hospital & Research Centre, Riyadh
  - National Guard King Abdulaziz Medical City, Riyadh
  - King Fahad Medical City, Riyadh
- Wits Donald Gordon Clinical Trial Centre, Parktown, Johannesburg, South Africa
- South Korea (7):
  - Kyungpook National University Chilgok Hospital, Daegu
  - National Cancer Center, Goyang-si
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St Mary's Hospital, Seoul
- Spain (11):
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona, Sant Andreu de la Barca, Barcelona
  - Complejo Hospitalario Universitario de Santiago (CHUS), Santiago de Compostela, LA Coruna
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Hospital Clínic i Provincial, Barcelona
  - Hospital Universitario Clínico San Cecilio, Granada
  - Hospital Juan Ramon Jimenez, Huelva
  - Centro Oncologico MD Anderson Internacional, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Hospital Arnau de Vilanova (Valencia) Servicio de Oncologia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (5):
  - Changhua Christian Hospital, Changhua
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital Office of General Surgery, Taipei
- Thailand (4):
  - Rajavithi Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Songklanagarind Hospital, Songkhla
- Turkey (Türkiye) (18):
  - Adana Baskent University Hospital, Adana
  - Ankara Oncology Hospital, Ankara
  - Gazi Uni Medical Faculty Hospital, Ankara
  - Ankara City Hospital, Ankara
  - Dicle University Faculty of Medicine, Diyarbakır
  - Trakya Universitesi Tip Fakultesi, Medikal Onkoloji Bilim Dali, Balkan Yerleskesi, Edirne
  - Ataturk University Medical Faculty Yakutiye Research Hospital Medical Oncology Department, Erzurum
  - Prof. Dr. Cemil Tascioglu City Hospital, Istanbul
  - Ac?badem Altunizade Hastanesi, Istanbul
  - Ege Uni Medical Faculty, Izmir
  - Katip Celebi University Ataturk Training and Research Hospital, Izmir
  - Kocaeli University Faculty of Medicine, İzmit
  - Erciyes Uni, Kayseri
  - Antalya Memorial Hastanesi, Kepez
  - Mersin City Education and Research Hospital, Mersin
  - Ondokuz Mayis Univ. Med. Fac., Samsun
  - Medical Park Seyhan Hospital, Seyhan
  - Namik Kemal Universitesi Tip Fakultesi, Medikal Onkoloji Bilim Dali, 100, Tekirdağ
- Uganda Cancer Institute, Kampala, Uganda
- United Arab Emirates (2):
  - Burjeel Medical City-Abu Dhabi, Abu Dhabi
  - Tawam Hospital, Al Ain City
- United Kingdom (11):
  - Ysbyty Gwynedd Hospital, Bangor
  - Royal United Hospital, Bath
  - Blackpool Victoria Hospital, Blackpool
  - University Hospital North Tees, Cleveland
  - Charing Cross Hospital, London
  - Maidstone Hospital, Maidstone
  - Nottingham University Hospitals NHS Trust - City Hospital, Nottingham
  - Royal Preston Hosp, Preston
  - North Wales Cancer Treatment Centre, Glan Clwyd Hospital, Rhyl
  - Singleton Hospital, Swansea
  - Royal Cornwall Hospital, Truro

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Kuemmel S, Harper-Wynne C, Park YH, Franke F, de Laurentiis M, Schumacher-Wulf E, Eiger D, Heeson S, Cardona A, Ozyilkan O, Morales-Vasquez F, Metcalfe C, Hafner M, Restuccia E, O'Shaughnessy J. heredERA Breast Cancer: a phase III, randomized, open-label study evaluating the efficacy and safety of giredestrant plus the fixed-dose combination of pertuzumab and trastuzumab for subcutaneous injection in patients with previously untreated HER2-positive, estrogen receptor-positive locally advanced or metastatic breast cancer. BMC Cancer. 2024 May 24;24(1):641. doi: 10.1186/s12885-024-12179-9. PMID 38789924